CLINICAL TRIAL: NCT07110298
Title: Association Between Angiography-based Quantitative Blood Flow Ratio and Peri-procedural Myocardial Injury：a Cohort Study
Brief Title: Association Between Peri-procedural Myocardial Injury and Quantitative Blood Flow Ratio
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: QFR AND PMI
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Coronary Arterial Disease (CAD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- post- procedural serum hs-cTNI level more than three times of URL: cohort divided into two groups based on the post- procedural serum hs-cTNI level

SUMMARY:
to apply angiography-based quantitative blood flow ratio to quantify the severity of the stenosed coronary artery prior to percutaneous coronary intervention, and monitor per-procedural myocardial injury based on the troponin level.Finally, to find the relationship between quantitative blood flow ratio results and myocardial injury degree.

ELIGIBILITY:
Inclusion Criteria:

* unstable angina patients

Exclusion Criteria:

* (1) multivessel diseases needed to be bypassed; (2) no track of high-sensitivity troponin I (hs-CTNI) level after PCI; (3) the elevated hs-CTNI level before PCI; (4) patients refusal to PCI; (5) side branch occlusion after PCI; (6) PCI failure with the main vessels occlusion; (7) eGRF (estimated glomerular filtration rate) less than 30ml/min/1.73m2; (8) no acquisition of QFR results because of the non-ideal angiographic quality.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: unstable angian patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
cardiovascular adverse events | three months
Major cardiac adverse events | three months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nienhuis MB, Ottervanger JP, Bilo HJ, Dikkeschei BD, Zijlstra F. Prognostic value of troponin after elective percutaneous coronary intervention: A meta-analysis. Catheter Cardiovasc Interv. 2008 Feb 15;71(3):318-24. doi: 10.1002/ccd.21345. PMID 18288753